CLINICAL TRIAL: NCT07240558
Title: Pandemic Influenza Vaccine in Organ Transplantation (PIVOT Trial): Safety and Immunogenicity of Pandemic Influenza Vaccine in Organ Transplant Recipients
Brief Title: Pandemic Influenza Vaccine in Organ Transplantation (PIVOT Trial)
Acronym: PIVOT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, Victoria Hall, Dr Victoria Hall, Principal Investigator, Clinician-Investigator and Infectious Diseases physician, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TID-2024-002; 196762 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Influenza (Pandemic); Avian Influenza; Vaccination
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — arepanrix; halofantrine

STUDY DESIGN:
Intervention Model Description: Randomized, placebo control trial 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- H5N1 vaccine (Active Comparator): This arm will receive 2 doses of approved H5N1 vaccine, 3 weeks apart
  Interventions: Biological: H5N1 vaccine (Arepanrix, GSK)
- Placebo (Placebo Comparator): This arm will receive 2 doses of normal saline (placebo), 3 weeks apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: H5N1 vaccine (Arepanrix, GSK) — 2 doses of H5N1 vaccine, 3 weeks apart, given IM (deltoid)
  Arms: H5N1 vaccine
Biological: Placebo — 2 doses of 0.5mls normal saline, 3 weeks apart, given IM (deltoid)
  Arms: Placebo

SUMMARY:
Influenza is an important pathogen in transplant recipients. The current widespread outbreak of highly pathogenic H5N1 avian influenza (HPAI) in livestock, and the occurrence of several human cases of infection suggest that the next influenza pandemic may be soon approaching. Transplant patients will likely be uniquely predisposed to serious infection with high morbidity and mortality. There are a number of important reasons that evaluation of prevention strategies are critical in this highly vulnerable population. Currently, there is no data on the immunogenicity of H5Nx vaccines in this highly vulnerable population. The investigators plan to study the safety and immunogenicity of a two-dose regimen of the pandemic influenza H5N1 vaccine in organ transplant patients.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double-blind, single-centre trial will evaluate the immunogenicity and safety of a two-dose regimen of the AS03-adjuvanted inactivated H5N1 vaccine (AREPANRIX™ H5N1, GSK) in adult organ transplant recipients. A total of 120 stable outpatient organ transplant recipients at the University Health Network (Toronto, Canada) will be enrolled and randomized 1:1 to receive two doses of H5N1 vaccine or placebo (0.9% saline) administered intramuscularly 3 weeks apart.

Blood samples collected at baseline (V0), 3 weeks (V1), and 6 weeks (V2) will be analyzed for serologic responses using hemagglutination inhibition (HAI) assays against vaccine and circulating H5N1 strains. In a subset of 60 participants (30 per arm), peripheral blood mononuclear cells will be obtained at each time point to assess cell-mediated immunity, including H5-specific CD4+ and CD8+ T-cell cytokine responses and B-cell immunity.

Participants will be monitored for local and systemic adverse events for 7 days following each dose and followed for 6 months for any adverse events, including rejection, influenza-like illness, and laboratory-confirmed influenza. Long-term immunogenicity will also be assessed at 6 months in vaccine recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and greater than 3 months post-transplant
* Stable graft function
* eGFR >30mL/min/1.73m2
* Able to provide informed consent

Exclusion Criteria:

* Allergy to vaccine components;
* Previous life-threatening reaction to influenza vaccine (ie Guillain Barré Syndrome);
* Ongoing or recent therapy for acute rejection (within the previous 30 days);
* Ongoing active cytomegalovirus (CMV) infection with viral load of greater or equal to 1000 international units/ml in the last 7 days;
* Febrile illness in the past 2 weeks;
* Rituximab in the last 6 months;
* Receiving treatment for active or acute infection;
* Unable to provide informed consent;
* 2025 seasonal influenza vaccination in preceding 6 weeks;
* Recent other vaccination in last 14 days;
* Receipt of intravenous immunoglobulin in last 30 days or expected to receive in next 30 days; Life expectancy < 3 months;
* Diagnosis of influenza virus infection in the last 90 days.
* Pregnancy known at the time of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Seroprotection and seroconversion 6 weeks after dose 1 | 6 weeks after dose 1 and 3 weeks after dose 2
  Participants with seroprotection (HAI titers greater than or equal to 1:40) after dose 2 AND seroconversion, defined as greater than or equal to 4-fold increase in HAI antibody titers from baseline to after dose 2 to the vaccine-matched H5 avian influenza strain.

SECONDARY OUTCOMES:
Seroprotection and seroconversion after dose 1 and comparison with after dose 2 | 6 weeks after dose 1
T and B cell immunity after dose 1 and dose of vaccine | 3 and 6 weeks post dose 1
Durability of immunity at 6 months post dose 1 | 6 months post dose 1
Local and systemic adverse events to vaccination | Until 6 months post dose 2
Other safety factors | Until 6 months post dose 2
  Transplant rejection, influenza like illness, confirmed influenza episodes
Seroprotection and seroconversion after dose 1 and 2 to H5, H1, H3 | 6 weeks and 3 weeks post dose 1

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Deidentified aggregated data will only be shared with appropriate request and ethical approval.